CLINICAL TRIAL: NCT01037153
Title: Effects of Nicotine on Brain Activity as Measured by fMRI
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999902371; 02-DA-N371
Record Dates: First submitted 2009-12-18; First posted 2009-12-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-07-25

CONDITIONS: Nicotine Dependence; Drug Abuse
Keywords: Intravenous; Rate of Delivery; Dose Responses; Variable Intervals; Multiple Rapid Injections
MeSH Terms: conditions — Tobacco Use Disorder; Substance-Related Disorders

SUMMARY:
Background:

- Nicotine addiction is common among people who smoke tobacco, and the addictive properties of nicotine make smoking cessation difficult even for people who want to quit. Research has shown that smoking causes changes in the brain that lead to addiction and craving, but more research is needed to determine how different doses of nicotine and different intervals of receiving nicotine affect brain function. A greater understanding of nicotine's effect on the brain, as studied through functional magnetic resonance imaging (fMRI), may improve the effectiveness of smoking cessation therapies and treatments.

Objectives:

- To determine the effects of nicotine on brain function and chemistry in experienced cigarette smokers.

Eligibility:

- Current smokers (at least 20 cigarettes per day for at least 1 year) between 18 and 50 years of age.

Design:

* The study involves five separate research experiments. Most participants will be involved in only one experiment.
* The experiments will evaluate brain activity and function using fMRI. Participants will be trained in a series of tests on cognitive function before beginning the experimental part of the study.
* Experiment 1: Participants will have three fMRI scan sessions after receiving different dose levels of intravenous nicotine.
* Experiment 2: Participants will have four fMRI scan sessions after receiving two doses of nicotine separated by 1/4, 1/2, 3, and 24 hours.
* Experiment 3: Participants will have two sets of nicotine injections separated by 45 minutes, with each injection series containing five rapid injections of small amounts of nicotine (to mimic five puffs on a cigarette).
* Experiment 4: Participants will have three fMRI sessions after receiving a single injection of nicotine at three different rates (over 15, 60, or 120 seconds). In addition there will be three more sessions involving a nicotine patch and a nicotine injection as well as a placebo session.
* Experiment 5: Participants will have three fMRI sessions that will involve looking at different kinds of pictures related to or not related to smoking after receiving a single injection of nicotine.
* Participants will also provide blood samples for further study....

DETAILED DESCRIPTION:
Objective:

The overall goal of this protocol is to employ fMRI to define nicotine's neural pharmacokinetic and pharmacodynamic properties and neurochemical sites and mechanisms of action in experienced smokers and to correlate these with monoamine and nicotinic receptor genotypes as well as to determine behavioral correlates of nicotine during various conditions of delivery and regress behavioral correlates of nicotine administration against neuroanatomical sites of activation across subjects.

Study Population:

The study population will consist of adult (18-50 y.o.) non-treatment seeking smokers. Subjects must smoke at least 20 cigarettes per day for at least 1 year. They cannot be dependent on any drug or alcohol except nicotine and caffeine. In addition, they must be appropriate candidates for fMRI scanning.

Design:

The study is divided into 5 separate arms with a maximum of two arms being conducted at one time. The experimental arms explore the effect of intravenous nicotine delivery with respect to the following parameters: dosage, interval of delivery, rate of delivery and emotional processing. Specifically the arms are as follows: Experiment 1: 3 fMRI scan sessions each administering either 0.25, 0.75 and 1.5 mg IV nicotine; Experiment 2: 4 fMRI scan sessions administering two doses of 1.25 mg nicotine separated by 0.25, 0.75, 3 and 24 hours; Experiment 3: two injection series separated by 45 minutes, each injection series containing 5 rapid injections of 0.25 mg each, much like 5 puffs on a cigarette; Experiment 4: 3 fMRI sessions administering a single injection of 1.5 mg nicotine at 3 different rates- over 15, 60 or 120 seconds; and Experiment 5: 3 fMRI session administering 1.5 mg nicotine followed by exposure to either neutral, negative, or positive affect pictures. Since experimental arms are conducted in series, rather than in parallel, there are very few subjects common to more than one experimental arm.

Outcome Measures:

The relevant outcome measures in this study are the behavioral and physiological effects and the patterns of brain regions activated (or suppressed) following the intravenous administration of nicotine across varying doses, intervals, rates and the effect on these parameters of emotional processing in the context of nicotine of stimuli with different affective valence.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Subjects must be between the ages of 18 - 50 and in good health, based on history and physical exam, and must demonstrate that they are experienced nicotine users based upon urine nicotine/cotinine levels or exhaled CO.
  2. Subjects must smoke a minimum of 20 cigarettes/day for at least 1 year.
  3. Subjects may be users of alcohol and/or marijuana but may not meet criteria for dependence on either and must have a negative urine drug triage prior to scanning.

EXCLUSION CRITERIA:

Subjects will be excluded if:

1. they are unable to undergo MRI scanning due to pregnancy, implanted metallic devices (cardiac pacemaker or neurostimulator, some artificial joints, metal pins, surgical clips or other implanted metal parts) or claustrophobia.
2. they have any major medical illnesses to include, but not limited to, hypertension, cardiovascular disease, asthma, diabetes, peripheral vascular diseases, coagulopathies, history of superficial or deep vein thrombosis, HIV, or other infectious diseases that may affect the CNS (e.g. syphilis).
3. they have any current major psychiatric disorders to include, but not limited to, mood, anxiety, psychotic disorders, or substance-induced psychiatric disorders.
4. they have history of neurological illnesses such as seizure disorders, migraine, multiple sclerosis, movement disorders, or history of head trauma, CVA, or CNS tumor.
5. they have alcohol or other drug dependence, other than nicotine dependence,
6. their T1 weighted brain MRI reveals gross structural abnormalities,
7. they have a history of syncope.
8. they are pregnant
9. they are actively seeking or engaged in smoking cessation treatment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Estimated)
Dates: Start 2002-08-06; Study Completion 2011-07-25

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute on Drug Abuse, Biomedical Research Center (BRC), Baltimore, Maryland, United States

REFERENCES:
- [Background] Aceto MD, Martin BR. Central actions of nicotine. Med Res Rev. 1982 Jan-Mar;2(1):43-62. doi: 10.1002/med.2610020104. No abstract available. PMID 6125634
- [Background] Avants SK, Margolin A, Kosten TR, Cooney NL. Differences between responders and nonresponders to cocaine cues in the laboratory. Addict Behav. 1995 Mar-Apr;20(2):215-24. doi: 10.1016/0306-4603(94)00066-2. PMID 7484315
- [Background] Bandettini PA, Jesmanowicz A, Wong EC, Hyde JS. Processing strategies for time-course data sets in functional MRI of the human brain. Magn Reson Med. 1993 Aug;30(2):161-73. doi: 10.1002/mrm.1910300204. PMID 8366797